CLINICAL TRIAL: NCT04008745
Title: Effect of Educational Booklet for Foot-related Exercises for Prevention and Treatment of Foot Musculoskeletal Dysfunctions of People With Diabetic Neuropathy: FOotCAre (FOCAtrial-II) Randomized Controlled Trial
Brief Title: Effect of Educational Booklet for Foot-related Exercises for Prevention and Treatment in People With Diabetic Neuropathy
Acronym: FOCA-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Isabel de Camargo Neves Sacco, Associate Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FOCA-II
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Neuropathies
Keywords: exercise therapy; diabetic foot; preventive care; foot-related exercise; self-management; musculoskeletal function; Booklet; Primary Health Care
MeSH Terms: conditions — Diabetic Neuropathies; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator (allocation, statistics, data processing) and assessor will be blid to the subjects allocation. To evaluate whether or not there was a failure in blinding of the outcome assessor, investigators and other assessors, they will be asked to guess which group the patients belonged to at the end of 8-weeks of treatment. Then the assessors will classify the certainty of their opinions according to a scale (1 = not sure, 5 = completely sure). To ensure that the assessor is not induced to correctly guess the participants' allocation, the patient will be instructed to not disclose any behavior details during the previous 8-weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients in the intervention group will perform foot-related exercises described in an educational booklet three times/week at home. In the follow-up period, patients will follow the same schedule set by the project till the end of the study (16-weeks).
  Interventions: Other: Educational and home-based physical therapy by foot-related exercises
- Control Group (No Intervention): Participants in the control group will not receive any specific intervention in addition to the treatment recommended by the health professionals team (doctors, nurses, podiatrists), which includes pharmacological treatment, and self-care recommendations and foot care by international consensus.

INTERVENTIONS:
Other: Educational and home-based physical therapy by foot-related exercises — The booklet is divided in 2: educational and exercise protocol. The aim of the first part is to guide the individual for a change in his/her health behavior, and comprises info about diabetic neuropathy, foot care, shoes, and benefits of exercising. The second part is the foot protocol, composed by 6 exercises. The maximum duration of a session is 20min and should be performed 3 times/week. The subject should warm-up the foot-ankle and then start exercising in the order suggested by the booklet, filling a table with the effort perceived (effort likert scale). The foot exercises progresses from one set with 30 repetitions in a sitting position, to exercising standing, then performing the exercise on one foot only. Other progression criterion is to increase the number of sets performed. The effort scale regulates the individual effort for his/her progression, which is also registered by the participant in the monthly table at the booklet.
  Arms: Intervention Group

SUMMARY:
The main objective of this trial is to investigate the effect of an educational booklet foot-related exercise in diabetic neuropathy status, functional outcomes and gait biomechanics in people with diabetic neuropathy.

DETAILED DESCRIPTION:
A randomized controlled trial will be performed with 48 patients with diabetic neuropathy. The participants will be randomly assigned into either a control group (recommended foot care by international consensus with no foot exercises) or an intervention group that will perform exercises at home, three times a week, through the booklet for 8-weeks.

The subjects will be evaluated in 3 different times to access the effect of the intervention: baseline and 8weeks, for all outcomes; and 16 weeks, for follow-up reasons for all outcomes.

The following outcomes will be assessed in all times: (1) diabetic neuropathy symptoms by Michigan Neuropathy Screening Instrument, (2) fuzzy score of the neuropathy severity, (3) tactile and vibration sensititivity (10-g monofilament and tuning fork), (4) foot-ankle kinematics and ankle kinetics during gait (infrared cameras and inverse dynamics, respectively), (5) foot isometric strength (by a pressure plate measurement), (6) functional balance reach test, (7) foot health and functionality by the Foot Health Status Questionnaire, (8) plantar pressure distribution during gait.

The hypothesis of this study is that the intervention will increase the perception of the tactile and vibratory sensitivity of the foot, reduce the symptoms of diabetic neuropathy, increase the strength of the foot muscles, increase the functional balance score, decrease the severity of the diabetic neuropathy (fuzzy score), decrease the number of neuropathy symptoms, promote a more physiological foot rollover with a redistribution of plantar pressure during gait, as well as increase foot-ankle mobility after 08-weeks of intervention. There will be also beneficial biomechanical changes during gait, such as: (1) increase in the ankle extensor moment and ankle concentric power in the propulsion phase and (3) increase in the ankle flexor moment and ankle eccentric power in the load phase.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 1 or 2;
* Moderate or severe neuropathy confirmed with the fuzzy software;
* Ability to walk independently in the laboratory

Exclusion Criteria:

* Hallux amputation or total amputation of the foot;
* History of surgical procedure in the knee, ankle or hip;
* History of arthroplasty and / or lower limb orthosis or indication of lower limb arthroplasty throughout the intervention period;
* Neurological and / or rheumatologic diseases diagnosed;
* Inability to provide consistent information;
* Perform physiotherapy intervention throughout the intervention period;
* Receiving any physiotherapy intervention or offloading devices;
* Major vascular complications;
* Severe retinopathy;
* Ulceration not healed for at least 6 months and / or active ulcer;
* Score between 12-21 (Probable Depression) from the Hospital Anxiety and Depression Scale (HADS).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel CN Sacco, PhD, Principal Investigator — Associate Professor at São Paulo University
Locations (1):
- Érica Queiroz da Silva, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silva EQ, Santos DP, Beteli RI, Monteiro RL, Ferreira JSSP, Cruvinel-Junior RH, Donini A, Verissimo JL, Suda EY, Sacco ICN. Feasibility of a home-based foot-ankle exercise programme for musculoskeletal dysfunctions in people with diabetes: randomised controlled FOotCAre (FOCA) Trial II. Sci Rep. 2021 Jun 11;11(1):12404. doi: 10.1038/s41598-021-91901-0. PMID 34117342
- [Derived] Silva EQ, Suda EY, Santos DP, Verissimo JL, Ferreira JSSP, Cruvinel Junior RH, Monteiro RL, Sartor CD, Sacco ICN. Effect of an educational booklet for prevention and treatment of foot musculoskeletal dysfunctions in people with diabetic neuropathy: the FOotCAre (FOCA) trial II, a study protocol of a randomized controlled trial. Trials. 2020 Feb 13;21(1):180. doi: 10.1186/s13063-020-4115-8. PMID 32054510
- See also: University of Sao Paulo website — http://www.usp.br
- See also: Laboratory of Biomechanics of Human Movement and Posture website — http://usp.br/labimph

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 25 | 25
Completed | 18 | 20
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (6.4) | 56.5 (9.4) | 57.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 6 | 5 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 25 | 25 | 50
Type 2 Diabetes [Count of Participants; unit: Participants] | 22 | 19 | 41
Time of onset of diabetes [Mean (Standard Deviation); unit: years] | 13.8 (10) | 18.2 (9.8) | 16 (9.9)
DPN symptoms - Michigan Neuropathy Screening Instrument [Mean (Standard Deviation); unit: score on a scale] — This questionnaire has 15 questions about the sensitivity of the feet and legs and is self-administered. A score of 1 point is given for answers of "yes" for questions 1, 2, 3, 5, 6, 8, 9, 11, 12, 14, and 15 and "no" for questions 7 and 13. Questions 4 and 10 evaluate circulatory deficits and general asthenia, respectively, and neither are included in the final score. The sum of all scores ranges from 0 to 13, and the larger the score, the worse the DPN.
  score on a scale | 5.4 (1.9) | 6.9 (2.1) | 6.2 (1.6)
Fuzzy classification of the DPN severity [Mean (Standard Deviation); unit: units on a scale] — The DPN severity will be made using the Decision Support System for Classification of Diabetic Polyneuropathy developed by the LaBIMPH. This decision will be based on fuzzy logic with the input variables of signs and symptoms extracted from the MNSI as well as tactile sensitivity (through the number of non-touch areas using a 10-g monofilament) and vibration sensitivity (by vibrating a tuning fork at 128 Hz), characterized as absent, present, or diminished. The software gives a score from 0 to 10, with higher scores indicating more severe DPN.
  units on a scale | 4.4 (2.6) | 4.9 (2.2) | 4.6 (2.4)
Body mass index (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 23.5 (4.8) | 22.9 (3.6) | 23.2 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Diabetic Neuropathy Symptoms at 8-weeks
Description: Score of the Michigan Neuropathy Screening Instrument (MNSI). This questionnaire comprises 15 questions about symptoms and events related to leg and foot sensitivity and is administered by the participant himself. The answers are summed to get a total score. The sum of all items results in a score ranging from 0 to 13 (13 represents the worst rating of the neuropathy).
Time Frame: 8-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
units on a scale | 5.3 (0.5) | 6.2 (0.6)

2. Primary Outcome: Change From Baseline of the Fuzzy Classification of the Diabetic Neuropathy Severity at 8-weeks
Description: The fuzzy classification of the diabetic neuropathy severity will be given by the Fuzzy software score developed by the Laboratory of Biomechanics of Movement and Human Posture (LaBIMPH) available free of charge at: http://www.usp.br/labimph/fuzzy/. It is a decision support system for classification of the diabetic neuropathy. This decision is based on three domains: signs and symptoms extracted from the Michigan Neuropathy Screening Instrument; tactile sensitivity through the number of non-sensible areas using a 10-g monofilament; and vibration sensitivity by vibrating a tuning fork (128Hz) characterized as absent, present or diminished. The software produces a score from 0 to 10 and the higher the score, the more severe the diabetic neuropathy.
Time Frame: 8-weeks
Measure: Mean (Standard Deviation); unit: score of a scale (0 to 10)
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
score of a scale (0 to 10) | 3.7 (0.5) | 3.3 (0.5)

3. Primary Outcome: Change From Baseline Diabetic Neuropathy Symptoms at 16-weeks (Follow-up)
Description: as for outcome 1
Time Frame: 16-weeks (Follow-up)
Measure: Mean (Standard Deviation); unit: score of a scale (0 to 13)
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
score of a scale (0 to 13) | 5.6 (0.5) | 6.0 (0.6)

4. Primary Outcome: Change From Baseline of the Fuzzy Classification of the Diabetic Neuropathy Severity at 16-weeks (Follow-up)
Description: as for outcome 2
Time Frame: 16-weeks (Follow-up)
Measure: Mean (Standard Deviation); unit: score of a scale (0 to 10)
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
score of a scale (0 to 10) | 3.9 (0.6) | 3.6 (0.4)

5. Secondary Outcome: Change From Baseline of the Foot and Ankle Kinematics During Gait at 8-weeks
Description: Sagital plane of ankle range of motion - initial of dorsiflexion until the end of plantaflexion (degrees) during stance phase of gait.
Time Frame: 8-weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
degrees | 23.7 (0.8) | 22.7 (0.8)

6. Secondary Outcome: Change From Baseline of the Foot and Ankle Kinetics During Gait at 8-weeks
Description: Peak joint moment of ankle plantarflexor moment at push off during stance phase of gait by inverse dynamic calculations
Time Frame: 8-weeks
Measure: Mean (Standard Deviation); unit: N*m/kg
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
N*m/kg | 1.3 (0.1) | 1.2 (0.1)

7. Secondary Outcome: Change From Baseline Dynamic Plantar Pressure Distribution During Gait at 8-weeks
Description: A pressure platform (emed®-q100, GmbH, Novel Munich, Germany) will be used to evaluate the pressure pattern during walking. The analysis of plantar pressure will be through the parameters: Heel peak pressure (kPa)
Time Frame: 8-weeks
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
kPa | 338.2 (19.0) | 402.4 (21.2)

8. Secondary Outcome: Change From Baseline Tactile Sensitivity at 8-weeks
Description: Tactile sensorial deficits will be evaluated by monofilament with a tactile stimulus of a 10-g monofilament in 4 plantar areas (plantar face of the hallux, heads of 1st, 3rd and 5th metatarsals). The areas will be evaluated in random order and not allowing the participant to view the monofilament. The number of areas where the participant does not feel the pressure will be indicated. The greater the number of areas marked without sensing, the greater the impairment of tactile sensitivity.
Time Frame: 8-weeks
Measure: Median (Inter-Quartile Range); unit: Number of insentitive foot areas
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 24
Number of insentitive foot areas | 0 [0 to 1] | 0 [0 to 2]

9. Secondary Outcome: Change From Baseline Vibration Sensitivity at 8-weeks
Description: The vibration sensitivity will be assessed by vibrating a tuning fork (128Hz) in the dorsal region of the distal hallux phalanx. The participant should report the moment he/she does no longer feel the vibration of the tuning fork, and the evaluator must time the interval between which the participant reports that he/she ceases to feel the vibration and the moment the evaluator ceases to feel the vibration in the his/her hand. Values smaller than 10 seconds will be classified with present vibratory sensitivity; values greater than 10 seconds will be classified as decreased vibratory sensitivity. If the participant does not perceive the vibration imposed by the tuning fork, it will be classified as absent vibratory sensitivity.
Time Frame: 8-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 23 | 20
Participants
  absent - L R | 12 | 11
  reduced - L R | 11 | 9

10. Secondary Outcome: Change From Baseline Foot Health and Functionality at 8-weeks
Description: The Brazilian version of the Foot-Health Status Questionnaire (FHSQ-BR) will be used. The domain assessed was function that receives a score from 0 to 100, where 100 expresses the best function and 0 to worst.
Time Frame: 8-weeks
Measure: Mean (Standard Deviation); unit: score on a scale (0 to 100)
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
score on a scale (0 to 100) | 37.0 (6.1) | 36.3 (5.1)

11. Secondary Outcome: Change From Baseline Foot Isometric Strength at 8-weeks
Description: The muscle strength of the flexor muscles of the hallux and flexors of the toes will be evaluated using the emed®-q100 pressure platform (Novel, Germany) according to a test protocol already described elsewhere. The individual should stand, with the evaluated foot centered on the pressure platform, instructed to make as much force as possible with the hallux peak values of maximum force (% of bodyweight).
Time Frame: 8-weeks
Measure: Mean (Standard Deviation); unit: % bodyweight
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
% bodyweight | 13.8 (1.1) | 11.6 (1.3)

12. Secondary Outcome: Change From Baseline Functional Balance at 8-weeks
Description: It is a clinical test where the patient will be standing barefoot, perpendicular to the wall, with the shoulder flexed 90° and the elbow extended. A tape measure will be attached to the wall, parallel to the floor, positioned at the height of the patient's acromion. The volunteer will be instructed to lean forward as much as possible without losing balance or taking a step. The displacement of the wrist will be measured by the tape. The greater the distance in centimeter, the better the functional balance
Time Frame: 8-weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
cm | 25.7 (1.3) | 25.5 (1.3)

13. Secondary Outcome: Change From Baseline of the Foot and Ankle Kinematics During Gait at 16-weeks (Follow-up)
Description: as for outcome 5
Time Frame: 16-weeks (Follow-up)
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
degrees | 24.6 (0.9) | 24.6 (0.8)

14. Secondary Outcome: Change From Baseline of the Foot and Ankle Kinetics During Gait at 16-weeks (Follow-up)
Description: Peak joint moment of ankle plantarflexor moment at push off during stance phase of gait by inverse dynamic calculations
Time Frame: 16-weeks (Follow-up)
Measure: Mean (Standard Deviation); unit: N*m/kg
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
N*m/kg | 1.20 (0.05) | 1.25 (0.03)

15. Secondary Outcome: Change From Baseline Dynamic Plantar Pressure Distribution During Gait at 16-weeks (Follow-up)
Description: as for outcome 7
Time Frame: 16-weeks (Follow-up)
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
kPa | 339.9 (15.7) | 378.4 (22.7)

16. Secondary Outcome: Change From Baseline Tactile Sensitivity at 16-weeks (Follow-up)
Description: as for outcome 8
Time Frame: 16-weeks (Follow-up)
Measure: Median (Inter-Quartile Range); unit: Number of insentitive foot areas
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
Number of insentitive foot areas | 0 [0 to 0] | 0 [0 to 1]

17. Secondary Outcome: Change From Baseline Vibration Sensitivity at 16-weeks (Follow-up)
Description: as for outcome 9
Time Frame: 16-weeks (follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 21 | 17
Participants
  absent - L R | 6 | 2
  reduced - L R | 15 | 15

18. Secondary Outcome: Change From Baseline Foot Health and Functionality at 16-weeks (Follow-up)
Description: The Brazilian version of the Foot-Health Status Questionnaire (FHSQ-BR) will be used. The domain assessed was function and it receives a score from 0 to 100, where 100 expresses the best function and 0 to worst.
Time Frame: 16-weeks (Follow-up)
Measure: Mean (Standard Deviation); unit: score on a scale (0 to 100)
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
score on a scale (0 to 100) | 40.3 (4.9) | 42.6 (6.2)

19. Secondary Outcome: Change From Baseline Foot Isometric Strength at 16-weeks (Follow-up)
Description: as for outcome 11
Time Frame: 16-weeks (Follow-up)
Measure: Mean (Standard Deviation); unit: % bodyweight
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
% bodyweight | 13.1 (1.3) | 12.0 (1.2)

20. Secondary Outcome: Change From Baseline Functional Balance at 16-weeks (Follow-up)
Description: as for outcome 12
Time Frame: 16-weeks (Follow-up)
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
cm | 26.0 (1.1) | 22.9 (1.1)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: The patients were advised to report any discomfort and foot pre-ulcerative signs (blisters, calluses) or foot ulcers to Researcher 3, who will ask for the blinded podiatrist nurse to assist the patient.
Groups:
- Intervention Group; Control Group: No adverse events were reported in relation to the intervention
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
It was a relatively short intervention period for major musculoskeletal and biomechanical changes, there was limited control over the exercise intensity, and only six exercises were included in the booklet. The participants were not blinded to the treatment. Control of glycated hemoglobin and glycemia. The education level of the participant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT04008745/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT04008745/ICF_001.pdf